CLINICAL TRIAL: NCT06051266
Title: Clinical Accuracy Evaluation of Dynamic Navigation and Static Template for Dental Implant Placement in Completely Edentulous Patients: A Randomized Parallel Controlled Multicenter Clinical Trial
Brief Title: Accuracy of Dynamic Navigation and Static Template in Completely Edentulous Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SDC-23-2
Record Dates: First submitted 2023-09-03; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-08

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic navigation (Experimental)
  Interventions: Device: Dynamic navigation
- Static template (Active Comparator)
  Interventions: Device: Static template

INTERVENTIONS:
Device: Dynamic navigation — Dynamic navigation eliminates the need for a laboratory fabrication process and allows for direct visualisation of the operative area during implant placement. Moreover, it can avoid interfering with water cooling. Navigation-assisted surgery makes it possible to modify the implant system, length, diameter or position in real time, both in the perioperative period and during surgery.
  Arms: Dynamic navigation
Device: Static template — In most clinical situations, a static template can be used to assist in guiding the placement of implants precisely. The static guide has some limitations in that it requires additional fabrication time, has insufficient cooling in the surgical field and is not suitable for simultaneous grafting procedures.
  Arms: Static template

SUMMARY:
The study was a prospective, multicentre, randomized parallel controlled clinical trial. Randomisation was conducted by central randomisation, with random allocation codes generated by the main central computer. Enrollment was conducted by competition between different centres. In this study, the coronal, apical and angular deviations (mean, standard deviation, median, quartiles, minimum, maximum, 95% confidence interval) of the static template and dynamic navigation group guided implant placement were calculated. The data is proposed to be analysed using a mixed linear effects model.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* American society of anesthesiologists (ASA) Levels 1 and 2
* Satisfy any of the following requirements:

  1. Edentulous maxillary patients
  2. Edentulous mandibular patients
  3. Terminally edentulous maxillary patients (number of remaining natural teeth in the upper jaw 1-4)
  4. Terminally edentulous mandibular patients (number of remaining natural teeth in the lower jaw 1-4)
  5. Full-mouth edentulous patients
  6. Full-mouth terminally edentulous patients (number of remaining natural teeth in one jaw 1-4)
* Implant-supported fixed restorations or implant-supported overdenture restorations
* Sufficient usable bone volume at implant sites, non-implant sites (≥1.5mm of remaining bone width on the labial/buccal and palatal/lingual sides after virtual implant placement in software)
* Maxillary and mandibular options for full-mouth patients are based on the inclusion of more single jaws in the non-bone grafted sites (see virtual peri-implant bone volume requirements in the pre-operative preparation phase)
* Mouth opening of 3 fingers or more
* Single-jawed missing patients treated with systemic periodontal therapy

Exclusion Criteria:

* Have a systemic disease that may affect prognosis (e.g. diabetic patients with glycated haemoglobin >6.5%, patients on bisphosphonate medication, patients with auto-systemic immune diseases, etc.)
* ASA grades 3 and 4
* Acute inflammation in the oral cavity: including uncontrolled periodontitis (periodontal probing depth > 4 mm) and untreated acute and chronic apical periodontitis
* Pregnancy or breastfeeding
* History of radiotherapy to the head and neck
* Heavy smokers (more than 10 cigarettes per day)
* Restricted mouth opening (less than three fingers).
* Participation in a clinical trial with another drug or device within 30 days prior to the start of the procedure (study day 0).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Apical deviation of implant placement (mm) | About 3 days after surgery
  Preoperative planning and postoperative cone-beam computed tomography (CBCT) were aligned together in the software and apical deviations(mm) of implant placement were measured to compare the results of the two groups.

SECONDARY OUTCOMES:
Coronal deviation of implant placement (mm) | About 3 days after surgery
  Preoperative planning and postoperative CBCT were aligned together in the software and coronal deviations(mm) of implant placement were measured to compare the results of the two groups.
Angular deviation of implant placement (°) | About 3 days after surgery
  Preoperative planning and postoperative CBCT were aligned together in the software and angular deviations(°) of implant placement were measured to compare the results of the two groups.
Operation time | Surgery day
  From anaesthesia to all implants are placed
Implant stability quotient | Surgery day
  Implant stability quotient was measured with the Osstell®device
visual analogue scale | About 3 days after surgery
  Patients were asked how they felt about the procedure using a visual analogue scale (VAS), which was measured using a visual analogue scale from 0 to 10. On a scale of 0 to 10 ("no pain" 0 to "maximum pain" 10) ("very comfortable" 0 to "not at all comfortable" 10) ("no swelling" 0 to "severe swelling" 10)
Failure rate | About 4 months after surgery
  Failure rate of implants during the healing period
Change of marginal bone level(mm) | About 1 year after surgery
  Marginal bone level = Measurement of the distance (mm) between the reference point (shoulder of the implant) and the point of bone-implant contact on the periapical film ; Change of marginal bone level = marginal bone level in the follow-up period - marginal bone level in the baseline period (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Yiqun Wu, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China